CLINICAL TRIAL: NCT01985100
Title: Hyperbaric Oxygen in the Reduction of Post Stroke Ischemic Penumbra
Brief Title: The Use of Hyperbaric Oxygen to Increase the Blood Supply in the Injured, But Still Alive Tissue, Around an Old Stroke
Acronym: HBO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit any patients that fulfilled the narrow enrollment requirements
Sponsor: John Davidson (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, John Davidson, Principal Investigator, St. Luke's Hospital, Chesterfield, Missouri
Organization: St. Luke's Hospital, Chesterfield, Missouri (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StLukesMO # 2013.021
Record Dates: First submitted 2013-11-07; First posted 2013-11-15 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single group (Experimental): single group of 6 patients will be treated with hyperbaric oxygen at 2 atmospheres absolute (ATA) for 90 minutes 5 days per week for 4 weeks (20 treatments) to see if the previously reported increase in cell metabolism following such treatment can be better documented by the more sensitive and precise method for assessing this, i.e. PET/MRI, than the previously reported SPECT/CT method
  Interventions: Other: hyperbaric oxygen chamber

INTERVENTIONS:
Other: hyperbaric oxygen chamber

SUMMARY:
To confirm or refute recently published data regarding the reduction in post-stroke ischemic penumbra, that used SPECT/CT, by using the more precise tools of PET/MRI.

DETAILED DESCRIPTION:
Most patients who suffer an acute ischemic stroke improve over the immediately ensuing 30-90 days. However, many patients do not improve beyond this initial period in spite of continued intensive physical therapy and supportive care. A prospective, randomized trial of the use of hyperbaric oxygen treatments in 59 such patients was published in January 2012. That study which used 40 hyperbaric oxygen treatments, indicated significant clinical neurological improvement in residual motor deficit in patients who had sustained a stroke over a year previously. An increase in brain activity in the region immediately surrounding their stroke (penumbra) was reported on the basis of SPECT studies. Regions of live cells were determined by CT. Because SPECT is primarily a measure of perfusion and not metabolic activity and CT is a poor measure of cell life, the investigators plan to assess areas of physiologic/anatomic mismatch in similar patients following hyperbaric oxygen treatment by the use of the more appropriate and precise tools, PET and MRI.

ELIGIBILITY:
Inclusion Criteria:

* person must have sustained an acute ischemic stroke 6-12 months prior to enrollment, exhibited clinical improvement during the initial 30-90 days post stroke, exhibited no further improvement for at least 1 month in spite of continued supportive care and physical therapy, must have at least one residual measurable motor deficit.

Exclusion Criteria:

Smoking, Contraindications to an MRI e.g. pacemaker, Contraindications to hyperbaric oxygen treatment e.g. emphysema, claustrophobia. seizure disorder, Inability to tolerate pressurization e.g. Eustachian tube dysfunction, other uncontrolled co-morbidities e.g. diabetes, hypertension, thyroid disorders, renal or hepatic dysfunction.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2014-09-27 (Actual); Study Completion 2014-09-27 (Actual)

PRIMARY OUTCOMES:
Increase in cellular metabolic activity in ischemic post stroke-penumbra PET scans | 2 weeks after treatment with Hyperbaric Oxygen

SECONDARY OUTCOMES:
Change in the motor function deficit post-stroke by Physical Therapists' measurements of motor strength | 2 weeks after completion of hyperbaric oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: John D Davidson, MD, Principal Investigator — St. Luke's Hospital St. Louis
Locations (1):
- St. Luke's Hospital, Chesterfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No